CLINICAL TRIAL: NCT06663878
Title: An Open-Label, Dose Escalation Study to Evaluate the Tolerability, Safety, and Preliminary Efficacy of MWAV201 in Subjects With Wilson Disease
Brief Title: An Exploratory Study to Evaluate the Tolerability and Safety of MWAV201 in Subjects With Wilson Disease
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Xinhua Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Collaborators: Mabwell (Shanghai) Bioscience Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MWAV201-CP101; 2021YFC2700802 (Other Grant/Funding Number: National Key Research and Development Program of China)
Record Dates: First submitted 2024-10-10; First posted 2024-10-29 (Actual); Last update posted 2024-10-29 (Actual); Status verified 2024-10

CONDITIONS: Wilson Disease
MeSH Terms: conditions — Hepatolenticular Degeneration

STUDY DESIGN:
Intervention Model Description: Participants will receive a single, peripheral intravenous (IV) infusion of MWAV201.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- MWAV201 (Experimental): All subjects will receive a single intravenous (IV) infusion of MWAV201.
  Interventions: Genetic: MWAV201

INTERVENTIONS:
Genetic: MWAV201 — Nonreplicating, recombinant gene transfer vector

SUMMARY:
The primary objective of this study is to evaluate the tolerability and safety of MWAV201 in patients with Wilson disease.

DETAILED DESCRIPTION:
This is an open-label, dose escalation study to evaluate the tolerability, safety, and preliminary efficacy of MWAV201 in patients with Wilson disease. Participants will receive a single, peripheral intravenous (IV) infusion of MWAV201. The dose escalation plan and the number of dose levels may be adjusted during study period.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged 18 and 65 years inclusive;
* Confirmed diagnosis of Wilson disease;
* Low copper diet and standardized medication for ≥ 1 year;
* Stable Wilson disease for ≥ 1 year;
* Able to understand and willing to follow study procedures.

Exclusion Criteria:

* Significant hepatic inflammation as evidenced by liver function test.
* Liver biopsy or liver stiffness measurement show progressive liver fibrosis.
* Laboratory tests or clinical symptoms indicate decreased liver reserve function.
* Other chronic liver disease (such as hepatitis B).
* Any signs of decompensated liver function (such as ascites).
* History of liver transplant or plan to receive liver transplant.
* Other diseases with clinical significance, such as cardiovascular and cerebrovascular diseases, kidney diseases, respiratory system diseases, neurological diseases, mental illnesses, active infections, etc.
* Body Mass Index ≥ 30 kg/m2.
* Other conditions that, in the Investigator's opinion, may not be suitable for the subject to be enrolled.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Estimated)
Dates: Start 2024-10 (Estimated); Primary Completion 2026-03 (Estimated); Study Completion 2031-05 (Estimated)

PRIMARY OUTCOMES:
Safety and tolerability profile [including adverse events (AEs) and serious adverse events (SAEs)] | At 1-Year post treatment
  AEs will be summarized based on incidence and the date of onset for the event.

SECONDARY OUTCOMES:
A Laboratory Outcome Measure: Total serum copper | At 1-Year post treatment
  Total serum copper will be summarized descriptively for all patients by dose cohort and planned visit, for absolute values, changes from baseline and percent change from baseline.
A Laboratory Outcome Measure: 24-hour urinary copper | At 1-Year post treatment
  24-hour urinary copper will be summarized descriptively for all patients by dose cohort and planned visit, for absolute values, changes from baseline and percent change from baseline.
A Laboratory Outcome Measure: Aspartate aminotransferase to platelet ratio index | At 1-Year post treatment
  Aspartate aminotransferase to platelet ratio index will be summarized descriptively for all patients by dose cohort and planned visit, for absolute values, changes from baseline and percent change from baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Jian-Gao Fan, doctor, Principal Investigator — Xinhua Hospital, Shanghai Jiao Tong University School of Medicine
Locations (1):
- Xinhua Hospital, Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No
This is a study initiated by investigator.